CLINICAL TRIAL: NCT05333627
Title: Internet-delivered Cognitive Behaviour Therapy for Post-Secondary Students: Preference Trial for Flexible, 5-Week, and 8-Week Options
Brief Title: Internet-delivered Cognitive Behaviour Therapy for Students: Duration Preference Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Ministry of Health, Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-205b
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Depression; Anxiety
Keywords: anxiety; depression; post-secondary students; internet-delivered cognitive behaviour therapy; transdiagnostic; preference trial
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Each client will choose one of the following: Wellbeing Course for Students (Fast-Track), Wellbeing Course for Students (5 weeks), and Wellbeing Course (8 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fast-Track Course (Experimental): Clients who select the Fast-Track Course option will receive access to a single ICBT core lesson and Do-It-Yourself guide, followed by three additional Do-It-Yourself guides that they can access in any order. The content includes examples that are tailored to students' experiences. Clients have access to diverse additional resources (e.g., managing panic, assertive communication) throughout the course. Clients will receive up to five weeks of optional therapist support.
  Interventions: Behavioral: Wellbeing Course for Students (Fast Track)
- 5-Week Course (Experimental): Clients who select the 5-week course will receive access to an ICBT course which consists of four lessons spread across the span of five weeks. The content includes examples that are tailored to students' experiences. Clients have access to diverse additional resources (e.g., managing panic, assertive communication) throughout the course. Clients will receive five weeks of optional therapist support.
  Interventions: Behavioral: Wellbeing Course for Students (5 weeks)
- 8-Week Course (Experimental): Clients who select the 8-week course will receive access to an ICBT course which consists of five lessons spread across the span of eight weeks. The content in this course is not student-specific. Clients have access to diverse additional resources (e.g., managing panic, assertive communication) throughout the course. Clients will receive eight weeks of optional therapist support.
  Interventions: Behavioral: Wellbeing Course (8 weeks)

INTERVENTIONS:
Behavioral: Wellbeing Course for Students (Fast Track) — The core Fast-Track lesson includes information on managing their cycle of symptoms, motivation, and an overview of strategies that can be used to manage symptoms of depression and anxiety. After the core lesson, clients can access three additional Do-It-Yourself guides that focus on thought challenging, controlled breathing/activity planning, and behavioural activation/relapse prevention. These materials are able to be accessed out of sequence on a schedule that suits their needs. With optional therapist support, therapists will respond to any messages that clients send once per week. Therapists will not message clients on weeks where the client does not send a message.
  Arms: Fast-Track Course
Behavioral: Wellbeing Course for Students (5 weeks) — The 5-week course consists of four lessons that provide psychoeducation about: symptom identification and the cognitive behavioural model, thought monitoring and challenging, controlled breathing and pleasant activity scheduling, graded exposure, and relapse prevention. With optional therapist support, therapists will respond to any messages that clients send once per week. Therapists will not message clients on weeks where the client does not send a message.
  Arms: 5-Week Course
Behavioral: Wellbeing Course (8 weeks) — The 8-week course consists of five lessons that provide psychoeducation about: symptom identification and the cognitive behavioural model, thought monitoring and challenging, controlled breathing and pleasant activity scheduling, graded exposure, and relapse prevention. With optional therapist support, therapists will respond to any messages that clients send once per week. Therapists will not message clients on weeks where the client does not send a message.
  Arms: 8-Week Course

SUMMARY:
There is growing evidence for the effectiveness of internet-delivered cognitive behaviour therapy (ICBT) for post-secondary students with symptoms of depression and anxiety. In ICBT, clients review structured online content over several weeks to learn strategies and skills to manage their symptoms. Low treatment completion rates remain a concern for post-secondary students, so it is possible that existing treatment protocols do not offer enough flexibility for students' needs and preferences.

This trial will examine students' preferences for different course options (fast-track, 5-week, and 8-week) and compare enrollment, adherence, and outcomes of students who pick each of the three options. In all three options, students will receive optional therapist support, in which the assigned therapist only contacts the student on weeks where the student sends the therapist a message. This trial will help inform the delivery of flexible treatment options for post-secondary students in a routine care setting.

ELIGIBILITY:
Inclusion Criteria:

* registered as a student at a post-secondary institution in Saskatchewan; over the age of 18; endorse symptoms of depression (score of 5 or greater on the PHQ-9) and/or anxiety (score of 5 or greater on the GAD-7); and be able to access computers and the Internet and be comfortable using them

Exclusion Criteria:

* high risk of suicide or hospitalization for mental health in previous 12 months; unmanaged alcohol or drug use problems; severe psychiatric illness that is not managed (e.g. psychosis or mania); or receiving other psychological services more than twice per month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | Baseline (screening), weeks 1-5 (Fast-Track and 5-week course), weeks 1-8 (8-week course), and week 16 (all course options)
  Change in depression symptoms. 9 items are summed into a total score, with scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (screening), weeks 1-5 (Fast-Track and 5-week course), weeks 1-8 (8-week course), and week 16 (all course options)
  Change in anxiety symptoms. 7 items are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.
Perceptions of Academic Functioning (PAF) | Baseline (screening), weeks 1-5 (Fast-Track and 5-week course), weeks 1-8 (8-week course), and week 16 (all course options)
  Change in subjective academic functioning. 3 items are summed into a total score ranging from 0 to 30, with higher scores indicating higher perceived functioning.

SECONDARY OUTCOMES:
Credibility and Expectancy Questionnaire (CEQ) | Baseline (screening), week 5 (Fast-Track and 5-week course), week 8 (8-week course)
  Measure of treatment credibility. Three items range from 0-9 with higher scores indicating better outcome.
Treatment Satisfaction | Week 5 (Fast-Track and 5-week course); Week 8 (8-week course)
  Measure includes 19 questions assessing satisfaction with various aspects of Internet-CBT and also negative effects of treatment
Work and Social Adjustment Scale (WSAS) | Baseline (screening), week 5 (Fast-Track and 5-week course), week 8 (8-week course)
  Measure includes 5 questions assessing impairment of functioning. Items are scored on a scale of 0 to 8. Total scores on the WSAS range from 0 to 40 with higher scores suggesting severe impairment.

OTHER OUTCOMES:
Alcohol Use Disorder Identification Test (AUDIT) | Baseline (screening)
  A 10-item screening tool to assess alcohol consumption. Items 1 to 8 are scored on a scale ranging from 0 to 4. Items 9 and 10 are scored on a three-point scale (0, 2, or 4). Scores from 10 items are summed with possible scores ranging from 0 to 40 and higher scores indicating a higher likelihood of problematic alcohol consumption.
Drug Use Disorder Identification Test (DUDIT) | Baseline (screening)
  An 11-item screening tool to assess problematic drug use. Items 1 to 9 are scored on a scale ranging from 0 to 4. Items 10 and 11 are scored as a 0, 2, or 4. Total scores for the DUDIT range from 0 to 44 with higher scores suggesting problematic drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Peynenburg, MA, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No